CLINICAL TRIAL: NCT01813838
Title: A Phase I-II Trial of Acadesine in IPSS High and Int-2 SMD, LAM With 20-30% Marrow Blasts and CMML Type 2 Not Responding to Azacitidine or Decitabine for at Least 6 Courses or Relapsing After a Response
Brief Title: GFM-Acadesine: A Phase I-II Trial of Acadesine
Acronym: Acadesine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Renal toxicity
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Advancell - Advanced In Vitro Cell Technologies, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003120-21
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2013-08

CONDITIONS: SMD
MeSH Terms: interventions — acadesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACADESINE 140mg/kg/d (Experimental): 3 patients will be included at the initial dose of Acadesine 140mg/kg/d
  Interventions: Drug: ACADESINE 140mg/kg/d
- ACADESINE 210mg/kg/d (Experimental): In absence of toxicity at the dose of 140mg/kg/d. There is a dose escalation of acadesine at the dose of 210mg/kg/d for 3 additionnal patients
  Interventions: Drug: ACADESINE 210mg/kg/d
- ACADESINE 315mg/kg/d (Experimental): In absence of toxicity at the dose of 210mg/kg/d. There is a dose escalation of acadesine at the dose of 315mg/kg/d for 3 additionnal patients
  Interventions: Drug: ACADESINE 315mg/kg/d

INTERVENTIONS:
Drug: ACADESINE 140mg/kg/d — 3 patients will be included at the initial dose of 140mg/kg/d. In absence of toxicity, 3 additional patients will be included at the higher dosage.
  In case of 1/3 toxicity, 3 additionnal patients will be included at the same dose level, currently 140mg/kg/d.
  In case of toxicity in 2 or more patients, the dose of acadesine will be reduced at the the dose of 85mg/kg/d
  Other Names: ACADESINE
  Arms: ACADESINE 140mg/kg/d
Drug: ACADESINE 210mg/kg/d — 3 patients will be included at the dose of 210mg/kg/d. In absence of toxicity, 3 additional patients will be included at the higher dosage.
  In case of 1/3 toxicity, 3 additionnal patients will be included at the same dose level, currently 210mg/kg/d.
  In case of toxicity in 2 or more patients, the dose of acadesine will be reduced at the the dose of 140mg/kg/d
  Other Names: ACADESINE
  Arms: ACADESINE 210mg/kg/d
Drug: ACADESINE 315mg/kg/d — 3 patients will be included at the dose of 315mg/kg/d.
  In case of 1/3 toxicity, 3 additionnal patients will be included at the same dose level, currently 315mg/kg/d.
  In case of toxicity in 2 or more patients, the dose of acadesine will be reduced at the the dose of 210mg/kg/d
  Other Names: ACADESINE
  Arms: ACADESINE 315mg/kg/d

SUMMARY:
A phase I-II trial of Acadesine in IPSS high and int 2 myelodysplastic syndromes, acute myeloid leukemia with 20-30% marrow blasts and chronic myelomonocytic leukemia type 2 not responding to Azacitidine or Decitabine for at least 6 courses or relapsing after a response:

Patients will receive 6 treatment cycles unless disease progression, transformation, or unacceptable toxicity occurs, or the patient refuses to continue participating in the study.

Efficacy will be assessed at the end of the 2nd, 4th and 6th cycles. After 6 cycles, patients demonstrating a response (CR, PR, marrow CR, or HI) will be able to continue with cycles of Acadesine (at the same dose as in the preceding cycles, depending on their cohort) until progression.

DETAILED DESCRIPTION:
Primary objectives

Phase I:

To determine the maximal tolerated dose (MTD) and dose limiting toxicities (DLTs) of increasing doses of IV Acadesine administered on D1, D3, D5, D8, D10 and D12 of 28 to 56 day-courses

Phase II:

To confirm safety and hematological toxicity in 18 additional patients

Secondary objectives:

Phase I:

* To determine response rates, as defined by the 2006 modified IWG criteria,
* To evaluate response duration, time to IPSS progression, and loss of RBC transfusion independence in these patients.
* To evaluate hospitalization duration, rates of rehospitalization for non-hematological toxicities, severe bleeding or febrile neutropenia.

Phase II:

To determine

* response rate as defined by the 2006 modified IWG criteria
* toxicity profile and safety
* response duration
* rate of progression to AML
* overall survival

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome including the following WHO categories: refractory anemia with excess blasts (RAEB), non-proliferative chronic myelomonocytic leukemia (CMML) (leukocytes < 13 G/L but > 10% marrow blasts), WHO- AML with 20-30% marrow blasts (RAEB-T according to the FAB classification)
* Prior treatment with Azacitidine or Decitabine for at least 6 courses without response (including CR, PR, marrow CR and stable disease with hematological improvement) or relapse after a response
* IPSS score >1 (IPSS: Int-2 or High);
* Age ≥ 18 years;
* Normal liver function tests, defined by total bilirubin and transaminases less than 1.5 time the upper limit of normal;
* Normal renal function, defined by creatinine less than 1.5 time the upper limit of normal, creatinine clearance ≥ 50 mL/min.
* Patient ineligible for allogeneic hematopoietic stem cell transplantation;
* Written informed consent;
* Patient must understand and voluntarily sign consent form;
* Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements;
* ECOG performance status between 0-2 at the time of screening;
* Women of childbearing potential must:

Agree to use effective contraception without interruption throughout the study and for a further 1 month after the end of treatment;

* Men must:

Agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and for a further 1 month after the end of treatment if their partner is of childbearing potential.

Exclusion Criteria:

* Severe infection or any other uncontrolled severe condition
* Significant cardiac disease - NYHA Class III or IV or having suffered a myocardial infarction in the last 6 months
* Less than 30 days since prior treatment with growth factors (EPO, G-CSF)
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
* Active cancer, or cancer during the year prior to trial entry other than basal cell carcinoma or carcinoma in situ of the cervix or breast;
* Patient already enrolled in another therapeutic trial of an investigational drug;
* HIV infection or active hepatitis B or C;
* Women who are or could become pregnant or who are currently breastfeeding;
* Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form;
* Patient eligible for allotransplantation.
* Known allergy to acadesine or any of its excipients
* No affiliation to an insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determine the maximal tolerated dose (MTD) | 6 month of treatment
  Phase I: Evaluation after 6 month of treatment. Responders will be treated until progression

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cluzeau, MD, Principal Investigator — Hôpital Saint Louis, Paris, France; Pierre Fenaux, MD, Principal Investigator — Hôpital Saint Louis, Paris, France
Locations (17):
- France (17):
  - Centre hospitalier de la côte Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU de Haut-Lévèque, Bordeaux Pessac
  - Centre henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Institut paoli calmettes, Marseille
  - centre hospitalier de Meaux, Meaux
  - CHU de nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital L'archet 1, Nice, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Centre henri Becquerel, Rouen
  - Hôpital Bretonneau de Tours, Tours

IPD SHARING:
Plan to Share IPD: No